CLINICAL TRIAL: NCT02218268
Title: Acute Effect of a Mixed Meal With and Without Extra Insulin on Arterial Stiffness, a Prospective Randomized Study.
Brief Title: Arterial Stiffness in Type I Diabetes Mellitus
Status: Completed | Type: Observational
Sponsor: University of Florida (Other)
Collaborators: Diabetes Action Research and Education Foundation (Other)
Responsible Party: Sponsor
Other Study IDs: IRB201400553; 00093792 (Other: University of Florida)
Record Dates: First submitted 2014-08-08; First posted 2014-08-18 (Estimated); Results first posted 2017-02-06 (Estimated); Last update posted 2017-02-06 (Estimated); Status verified 2016-12

CONDITIONS: Arterial Stiffness in Youth With Type 1 Diabetes
Keywords: type I diabetes; healthy; children; adolescents; young adults
MeSH Terms: conditions — Diabetes Mellitus, Type 1

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Pre-meal bolus then No meal bolus: A meal replacement drink (Boost) and bolus of rapid insulin will be given to this group. Glucose will be monitored with a finger prick before they drink the meal replacement, 1 hour later and finally 2 hours after drinking the meal replacement. Stiffness of the blood vessel of the wrist will be determined using radial tonometry and will be done at the same time as the glucose monitoring.
  Then 3 months later A meal replacement drink (Boost) will be given but the subject will not receive a meal bolus. Glucose will be monitored with a finger prick before they drink the meal replacement, 1 hour later and finally 2 hours after drinking the meal replacement. Stiffness of the blood vessel of the wrist will be determined using radial tonometry and will be done at the same time as the glucose monitoring
  Interventions: Drug: Pre-meal bolus; Drug: No meal bolus
- No meal bolus then Pre-meal bolus: A meal replacement drink (Boost) will be given but the subject will not receive a meal bolus. Glucose will be monitored with a finger prick before they drink the meal replacement, 1 hour later and finally 2 hours after drinking the meal replacement. Stiffness of the blood vessel of the wrist will be determined using radial tonometry and will be done at the same time as the glucose monitoring.
  Then 3 months later meal replacement drink (Boost) and bolus of rapid insulin will be given to this group. Glucose will be monitored with a finger prick before they drink the meal replacement, 1 hour later and finally 2 hours after drinking the meal replacement. Stiffness of the blood vessel of the wrist will be determined using radial tonometry and will be done at the same time as the glucose monitoring
  Interventions: Drug: Pre-meal bolus; Drug: No meal bolus

INTERVENTIONS:
Drug: Pre-meal bolus — Long acting insulin as scheduled per usual routine PLUS rapid/ short acting (bolus) prior to Boost
Drug: No meal bolus — Long Acting insulin as scheduled per usual routine (given once daily)

SUMMARY:
Using radial artery tonometry to study arterial stiffness, the plan is to study a cohort of 65 children with Type I diabetes mellitus. This prospective, crossover study will help determine if there is an acute increase in arterial stiffness in children with Type I diabetes mellitus who do not give extra insulin to cover a meal. This will give more support to show why it is so critical to bolus every time they eat and to bolus on time to decrease cardiovascular consequences of poorly controlled diabetes. The hypothesis is that giving insulin before a meal compared to not giving insulin before a meal will be associated with lower arterial stiffness in children with type I diabetes.

DETAILED DESCRIPTION:
The subject will fast overnight (nothing to eat or drink for at least 8 hours). The subject will be asked to drink a mixed meal replacement drink (Boost) and will be randomized (like flipping a coin) to bolus insulin for the "meal" or to not bolus insulin using their standard insulin dose. Glucose will be monitored with a finger prick before they drink the meal replacement, 1 hour later and finally 2 hours after drinking the meal replacement.

Stiffness of the blood vessel of the wrist will be determined using radial tonometry. Radial tonometry is safe and does not hurt. A pen like probe is placed on the blood vessel of the wrist. When the machine reads a good wave form the computer will calculate the stiffness of the blood vessel. This test will be done along with the glucose checks; before drinking the meal replacement drink, and 1 and 2 hours after drinking the meal replacement drink.

During the next study visit, the subject will repeat the exact same study described above. However, this time they will receive the other insulin assignment they were assigned during the first study (either bolus or no bolus).

ELIGIBILITY:
Inclusion Criteria:

* Type 1 diabetes based on clinical history
* Basal-bolus insulin regimen
* Duration of diabetes greater than 1 year
* Blood glucose 65-200 mg/dL fasting

Exclusion Criteria:

* Use of metformin or any other hypoglycemic agents besides insulin
* Use of anti-hypertensives
* Caffeine or smoking within the past 24 hours

Ages: 8 Years to 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: University of Florida diabetes clinic and the Florida Camp for Children and Youth with Diabetes. Subjects had type 1 diabetes for at least one year, were using a basal-bolus insulin regimen, and were not taking oral hypoglycemic agents or antihypertensive drugs.
Sampling Method: Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2014-10; Primary Completion 2015-08 (Actual); Study Completion 2015-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael Haller, MD, Principal Investigator — University of Florida
Locations (1):
- University of Florida, Gainesville, Florida, United States

RESULTS

PARTICIPANT FLOW:
Period: First Phase (2 Hours)
Arm/Group | Pre-meal Bolus Then No Meal Bolus | No Meal Bolus Then Pre-meal Bolus
Started | 30 | 30
Completed | 30 | 30
Not Completed | 0 | 0
Period: 24 Hour Washout
Arm/Group | Pre-meal Bolus Then No Meal Bolus | No Meal Bolus Then Pre-meal Bolus
Started | 30 | 30
Completed | 19 | 21
Not Completed | 11 | 9
Not completed — Physician Decision | 11 | 9
Period: Final Phase (2 Hours)
Arm/Group | Pre-meal Bolus Then No Meal Bolus | No Meal Bolus Then Pre-meal Bolus
Started | 19 | 21
Completed | 19 | 21
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- All Participants: This is a crossover study of youth with Diabetes on a stable basal bolus insulin regimen. They will be randomized either receive a pre-meal insulin bolus in conjunction with their Basal insulin bolus or receive their standard of care basal insulin bolus only. A mixed meal replacement (Boost) will be consumed. Glucose will be monitored with a finger prick before they drink the meal replacement, 1 hour later and finally 2 hours after drinking the meal replacement. Stiffness of the blood vessel of the wrist will be determined using radial tonometry and will be done at the same time as the glucose monitoring. This is a crossover study and all participants will take place in this arm after 3 months of their visit.
Arm/Group | All Participants
Number analyzed (Participants) | 60
Age, Continuous [Mean (Standard Deviation); unit: years] | 12.5 (2.13)
Gender [Count of Participants; unit: Participants]
  Female | 32
  Male | 28
Region of Enrollment [Number; unit: participants]
  United States | 60
HbA1c [Mean (Standard Deviation); unit: percentage] | 7.86 (0.96)

OUTCOME MEASURES:

1. Primary Outcome: Determine the Difference Between Acute Effect of a Mixed Meal on Radial Artery Stiffness in Subjects With Type I Diabetes Mellitus Who do and Who do Not Take an Additional Bolus of Insulin.
Description: Determine the difference between acute effect of a mixed meal on radial artery stiffness in subjects with type I diabetes mellitus who do and who do not take an additional bolus of insulin. Radial tonometry is used to calculate the augmentation index (AI). AI is expressed as a percentage of the pulse pressure and represents the difference between the first and second peaks of the central arterial waveform. The stiffer the artery the more positive elevation of the AI and the machine will indicate stiffness using a color indicator (green less stiff and red being stiff). AI is measured using the SphygmoCor VX version 7.01 (AtCor Medical, Syndey, Australia). AI will be corrected to a heart rate of 75 to eliminate differences related to heart rate variation.
Time Frame: From baseline to one hour then 2 hours
Measure: Mean (95% Confidence Interval); unit: Percent of Pulse Pressure
Arm/Group | Pre-meal Bolus Then No Meal Bolus | No Meal Bolus Then Pre-meal Bolus
Number analyzed (Participants) | 19 | 21
Percent of Pulse Pressure
  Difference of mean AI75 1 hour after | -4.5 [-7.97 to -1.1] | -4.5 [-7.97 to -1.1]
  Difference of mean AI75 2 hours after | -4.3 [-8.9 to 0.2] | -4.3 [-8.9 to 0.2]

ADVERSE EVENTS:
Groups:
- Pre-meal Bolus Then No Meal Bolus: A meal replacement drink (Boost) and bolus of rapid insulin will be given to this group. Glucose will be monitored with a finger prick before they drink the meal replacement, 1 hour later and finally 2 hours after drinking the meal replacement. Stiffness of the blood vessel of the wrist will be determined using radial tonometry and will be done at the same time as the glucose monitoring. This is a crossover study and all participants will take place in this arm after 3 months of their visit.
- No Meal Bolus Then Pre-meal Bolus: A meal replacement drink (Boost) will be given but the subject will not receive a meal bolus. Glucose will be monitored with a finger prick before they drink the meal replacement, 1 hour later and finally 2 hours after drinking the meal replacement. Stiffness of the blood vessel of the wrist will be determined using radial tonometry and will be done at the same time as the glucose monitoring, This is a crossover study and all participants will take place in this arm after 3 months of their visit.
Arm/Group | Pre-meal Bolus Then No Meal Bolus | No Meal Bolus Then Pre-meal Bolus
Serious Adverse Events (participants affected / at risk) | 0/30 | 0/30
Other Adverse Events (participants affected / at risk) | 0/30 | 0/30

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No